CLINICAL TRIAL: NCT04543994
Title: A Phase IB/IIA Study of Remestemcel-L, an ex Vivo Culture-expanded Adult Allogeneic Bone Marrow Derived Mesenchymal Stem Cell Product, for the Treatment of Medically Refractory Ulcerative Colitis
Brief Title: Study of Mesenchymal Stem Cells for the Treatment of Medically Refractory Ulcerative Colitis (UC)
Acronym: UC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cleveland Clinic (Other)
Collaborators: Mesoblast, Inc. (Industry)
Responsible Party: Principal Investigator, Amy Lightner, Principal Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-1005
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; medically refractory ulcerative colitis; UC; refractory ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — remestemcel-l

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Remestemcel-L (150 million cells) (Experimental): Targeted endoscopic delivery of remestemcel-L at a dose of 150 million cells into the submucosal layer of the colon wall at baseline.
  If at 3 months post injection of remestemcel-L there is clinical, endoscopic or radiographic improvement, patients will receive a second dose of remestemcel-L at a dose of 150 million MSCs (same dose at initial).
  Interventions: Drug: Remestemcel-L
- Remestemcel-L (300 million cells) (Experimental): Targeted endoscopic delivery of remestemcel-L at a dose of 300 million cells into the submucosal layer of the colon wall at baseline.
  If at 3 months post injection of remestemcel-L there is clinical, endoscopic or radiographic improvement, patients will receive a second dose of remestemcel-L at a dose of 300 million MSCs (same dose at initial).
  Interventions: Drug: Remestemcel-L
- Placebo (Placebo Comparator): Direct injection of normal saline into the submucosal layer of the colon wall.
  If not completely healed after 3 months, participants will then cross over to the treatment group to receive a direct injection of remestemcel-L at a dose of 150 or 300 million cells into the submucosal layer of the colon wall.
  If at 6 months post injection of remestemcel-L there is clinical, endoscopic or radiographic improvement, patients will receive a second dose of remestemcel-L at a dose of 150 or 300 million MSCs (same dose at initial).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Remestemcel-L — An ex vivo culture-expanded adult allogeneic bone marrow derived mesenchymal stem cell product for the treatment of medically refractory ulcerative colitis
  Arms: Remestemcel-L (150 million cells)
Drug: Remestemcel-L — An ex vivo culture-expanded adult allogeneic bone marrow derived mesenchymal stem cell product for the treatment of medically refractory ulcerative colitis
  Arms: Remestemcel-L (300 million cells)
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of using remestemcel-L, an ex vivo culture-expanded adult allogeneic bone marrow derived mesenchymal stem cell product (MSCs) delivered by targeted endoscopic delivery to treat people for medically refractory ulcerative colitis.

This study will enroll adult patients with medically refractory ulcerative colitis who are planning to switch biologic therapy or undergo colectomy as the next stage in their treatment plan.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is an idiopathic chronic inflammatory disease of the colon and rectum, which continues to increase in incidence for unknown reasons, resulting in a significant burden to the healthcare system. UC is characterized by persistent mucosal inflammation of the colon and rectum with a chronic remitting and relapsing behavior which leaves patients on chronic immunosuppression and hospitalizations to treat the disease symptoms, but unable to cure the disease. Despite the ever-growing armamentarium of immunosuppressive medication, up to 30% of patients still require a colectomy for medically refractory disease.

Participants with medically refractory ulcerative colitis will be treated by targeted endoscopic delivery of remestemcel-L, an ex vivo culture expanded allogeneic bone marrow derived mesenchymal stem cell product at a dose of 150 or 300 million. This will be injected into the submucosal layer of the colon and rectal wall.

Patients will receive a second dose of remestemcel-L at a dose of 150 or 300 million MSCs (same dose as initial). If at 3 months post injection of remestemcel-L there is clinical remission, escalation of medical management and/or surgery will be delayed and patients observed. If there is worsening or no improvement in treated patients, then patients will proceed with escalation of medical management or colectomy as per standard of care. Control patients without improvement will cross over to receive remestemcel-L at 3 months and may be retreated at 6 months. All patients will be followed for two years post initial treatment.

There will be a total of 4 cohorts of 3 patients (2 treatment:1 control) receiving the 150 million MSC dose of study drug and a total of 4 cohorts of 3 patients (2 treatment:1 control) receiving 300 million MSCs dose of study drug. This study plans to enroll a total of 24 participants.

The primary endpoint of this study is to determine the safety and feasibility of endoscopic injection of remestemcel-L, an ex vivo culture expanded allogeneic bone marrow derived mesenchymal stem cell product for treatment of medically refractory ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria

1. Males and Females 18-75 years of age.
2. Ulcerative colitis of at least 6 months duration with medically refractory symptoms
3. Exposure to corticosteroids, 5-ASA drugs, thiopurines, methotrexate, anti-TNF therapy, anti-integrin and anti-interleukin in the past are permitted but a washout period of 4 weeks for any monoclonal antibody is necessary.

   1. If receiving conventional immunomodulators (ie, AZA, 6-MP, or MTX), must have been taking them for ≥12 weeks, and on a stable dose for at least 4 weeks.
   2. If AZA, 6-MP, or MTX has been recently discontinued, it must have been stopped for at least 4 weeks.
   3. If receiving oral 5-ASA compounds, the dose must have been stable for at least 4 weeks.
   4. If receiving oral corticosteroids, the dose must be ≤20 mg/day prednisone or its equivalent and must have been stable for at least 4 weeks.
   5. If receiving budesonide, the dose must have been stable for at least 2 weeks.
   6. If oral 5-ASA compounds or oral corticosteroids (including budesonide) have been recently discontinued, they must have been stopped for at least 2 weeks.
4. The following medications/therapies must have been discontinued before first administration of study agent:

   1. TNF-antagonist therapy (eg, infliximab, etanercept, certolizumab, adalimumab, golimumab), vedolizumab, ustekinumab for at least 4 weeks.
   2. Cyclosporine, tacrolimus, or sirolimus, for at least 4 weeks.
   3. 6-thioguanine (6-TG) must have been discontinued for at least 4 weeks.
   4. Rectal corticosteroids (ie, corticosteroids [including budesonide] administered to the
   5. rectum or sigmoid colon via foam or enema or suppository) for at least 2 weeks.
   6. Rectal 5-ASA compounds (ie, 5-ASAs administered to the rectum or sigmoid colon viafoam or enema or suppository) for at least 2 weeks.
   7. Parenteral corticosteroids for at least 2 weeks.
   8. Total parenteral nutrition (TPN) for at least 2 weeks.
   9. Antibiotics for the treatment of UC (eg, ciprofloxacin, metronidazole, or rifaximin) for at least 2 weeks.
5. No colonic dysplasia and malignancy as ruled out by colonoscopy within 30 days of MSC delivery
6. Ability to comply with protocol
7. Competent and able to provide written informed consent
8. Must have lost response to at least one monoclonal antibody (anti-TNF, anti-interleukin, or anti-integrin therapy), tofacitinib, or have a contra-indication to biologic therapy
9. If patient is of reproductive capacity, willing to use adequate birth control measures while they are in the study

Exclusion Criteria for all patients to join the protocol

1. Inability to give informed consent.
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
3. Specific exclusions;

   1. HIV
   2. Hepatitis B or C
4. Abnormal AST or ALT at screening defined as AST >100 or ALT > 100
5. Abnormal basic laboratory values with the following cut-offs:

   1. Alkaline phosphate >200
   2. WBC >13
   3. Hemoglobin <7
   4. Platelets <50 or > 1 million
   5. Creatinine >1.5
6. History of cancer including melanoma (with the exception of localized skin cancers) within 5 years of study enrollment
7. Investigational drug within one year of study enrollment
8. Pregnant or breast feeding.
9. Fulminant colitis requiring emergency surgery
10. Concurrent active clostridium difficile infection of the colon
11. Concurrent CMV infection of the colon
12. Evidence of colonic perforation
13. Massive hemorrhage from the colon requiring emergent surgery
14. Crohn's colitis or indeterminate colitis
15. Microscopic, ischemic or infectious colitis
16. Neoplasia of the colon and preoperative biopsy
17. Presence of an ostomy
18. Prior small bowel resection
19. Previous colonic resection
20. Colonic stricture that unable to pass an adult colonoscope
21. Active or latent tuberculosis
22. Unable to wean off corticosteroids
23. Patients with extra colonic ulcerative colitis including primary sclerosing cholangitis
24. Patients with history of or current evidence of alcohol or drug abuse or dependence, recreational use of illicit drug or prescription medications, or have use of medical marijuana within 90 days of study entry
25. Patients with known allergy to local anesthetics
26. Patients with a known allergy to DMSO, porcine and/or bovine proteins
27. Patients taking anticoagulant medications (e.g. warfarin, heparin) or clopidogrel (Plavix) to reduce the risk of bleeding/ hemarthrosis
28. If patient is of reproductive capacity, unwilling to use adequate birth control measures while they are in the study

Control patients will have additional criteria that need to be met prior to the patients crossing over to receive treatment.

Inclusion Criteria for control patients prior to entering the treatment phase:

1. Received placebo at the point of first injection
2. Completed all study visits to date
3. Clinical status has remained the same or improved, not worsened

Exclusion Criteria for control patients who will be entering the treatment phase:

1. Required repeat hospitalization for a colitis flare
2. Given oral and intravenous steroids for a colitis flare
3. Had worsening abdominal pain frequency of bowel movements, blood in stool
4. Desires exclusion from the study to pursue escalation in medical management or surgery Allogeneic Bone
5. Has a colonic perforation that requires surgery
6. Has colonic bleeding that requires surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events | Month 3
  Number of participants with treatment related adverse events post-injection of 150 or 300 million allogeneic bone marrow derived mesenchymal stem cells for the treatment of medically refractory Ulcerative colitis as assessed by protocol CCF-Stem Cells IBD-005.

SECONDARY OUTCOMES:
Clinical and endoscopic remission | Month 3, Month 12
  Number of participants with clinical and endoscopic remission post-injection of 150 or 300 million bone marrow allogeneic derived mesenchymal stem cells for the treatment of medically refractory Ulcerative colitis.
  Clinical and endoscopic remission is defined as:
  Clinical remission: Mayo Clinic score of 2 or lower and no subscore higher than 1, and mucosal healing, defined as an endoscopic subscore of 0 or 1
  Endoscopic remission: Mayo Clinic scale endoscopic subscore of 0 or 1
Clinical and endoscopic response | Month 3, Month 12
  Number of participants with a clinical and endoscopic response post-injection of 150 or 300 million allogeneic bone marrow derived mesenchymal stem cells for the treatment of medically refractory Ulcerative colitis.
  Clinical and endoscopic response is defined as:
  Clinical response: Reduction in the Mayo Clinic score by 3 points and a decrease of at least 30% from the baseline score with a decrease of at least 2 points on the rectal bleeding subscale to an absolute rectal bleeding score of 1 or 2.
  Endoscopic response: Mayo Clinic scale endoscopic subscore decrease by at least one point
Partial clinical and endoscopic response | Month 3, Month 12
  Number of participants with a partial clinical and endoscopic response post-injection of 150 or 300 million allogeneic bone marrow derived mesenchymal stem cells for the treatment of medically refractory Ulcerative colitis.
  Partial clinical and endoscopic response is defined as:
  Partial clinical response: Reduction in the Mayo Clinic score that does not meet the following: by 3 points and a decrease of at least 30% from the baseline score with a decrease of at least 2 points on the rectal bleeding subscale to an absolute rectal bleeding score of 1 or 2
  Partial endoscopic response: No improvement in Mayo Clinic scale endoscopic subscore that stays the same or decreases
Lack of response | Month 3, Month 12
  Number of participants with a lack of response post-injection of 150 or 300 million allogeneic bone marrow derived mesenchymal stem cells for the treatment of medically refractory Ulcerative colitis.
  Lack of response is defined as:
  Clinical response: No improvement in Mayo Clinic score
  Endoscopic response: No improvement or worsening in Mayo Clinic scale endoscopic subscore
Mayo clinic score | Month 1 through Month 24
  Mayo clinic score will be used to measure quality of life in participants.
  *Score ranges from 0 (least severe) to 12(most severe).

OTHER OUTCOMES:
Inflammatory bowel disease questionnaire | Month 1 through Month 24
  Inflammatory bowel disease questionnaire will be used to measure quality of life in participants.
  *Score ranges from 32 (best health) to 224 (worst health)
EuroQol 5 Dimensions survey | Month 1 through Month 24
  EuroQol 5 Dimensions survey will be used to measure quality of life in participants.
  *Score ranges from 5 (full health) to 25 (worst health).
IBD-patient reported treatment impact survey | Month 1 through Month 24
  IBD-patient reported treatment impact survey will be used to measure quality of life in participants.
  *Score ranges from 3 (most satisfied) to 15 (least satisfied)
Short Form 36 health survey | Month 1 through Month 24
  Short Form 36 health survey will be used to measure quality of life in participants.
  *Score ranges from 0 (least favorable health state) to 3600 (most favorable health state)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lightner, Principal Investigator — Cleveland Clinic Foundation, Cleveland OH
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandborn WJ, Feagan BG, Rutgeerts P, Hanauer S, Colombel JF, Sands BE, Lukas M, Fedorak RN, Lee S, Bressler B, Fox I, Rosario M, Sankoh S, Xu J, Stephens K, Milch C, Parikh A; GEMINI 2 Study Group. Vedolizumab as induction and maintenance therapy for Crohn's disease. N Engl J Med. 2013 Aug 22;369(8):711-21. doi: 10.1056/NEJMoa1215739. PMID 23964933
- [Background] Kin C, Kate Bundorf M. As Infliximab Use for Ulcerative Colitis Has Increased, so Has the Rate of Surgical Resection. J Gastrointest Surg. 2017 Jul;21(7):1159-1165. doi: 10.1007/s11605-017-3431-0. Epub 2017 May 8. PMID 28484890